CLINICAL TRIAL: NCT02504814
Title: Physiological and Clinical Changes in NHF Therapy
Acronym: ATMOFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Jens Bräunlich, MD, MD, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 414-14-06102014
Record Dates: First submitted 2015-05-27; First posted 2015-07-22 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnia; Interstitital Lung Disease
Keywords: nasal high flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ventilatory effects (Experimental): measuring mean airway pressure, breathing volumes and decrease in hypercapnia
  Interventions: Device: Nasal Highflow (NHF)

INTERVENTIONS:
Device: Nasal Highflow (NHF) — changes in breathing physiology in NHF
  Other Names: TNI softflow50

SUMMARY:
The study explores the changes in pressure, volume and in hypercapnia in patients with COPD and ILD. The investigators will use different application forms.

ELIGIBILITY:
Inclusion Criteria:

* COPD, ILD

Exclusion Criteria:

* Unstable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
changes in mean airway pressure (mbar) | 1 month
changes in tidal and minute volume (l) | 1 month
changes in breathing frequency (beats/ minute) | 1 month

SECONDARY OUTCOMES:
changes in partial pressure of carbon dioxide (CO2) in arterial blood (pCO2) | 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bräunlich, MD, Study Director — University of Leipzig
Locations (1):
- Jens Bräunlich, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Braunlich J, Mauersberger F, Wirtz H. Effectiveness of nasal highflow in hypercapnic COPD patients is flow and leakage dependent. BMC Pulm Med. 2018 Jan 24;18(1):14. doi: 10.1186/s12890-018-0576-x. PMID 29368599